CLINICAL TRIAL: NCT05493267
Title: A Exploratory Study of Vγ2Vδ2 T Lymphocyte-based Immunotherapy for MDR-TB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Shanghai Public Health Clinical Center (Other Government); Huashan Hospital (Other); No.85 Hospital, Changning, Shanghai, China (Other)
Responsible Party: Principal Investigator, Wei Sha MD & PhD, Director, Head of Tuberculosis Department,Shanghai Pulmonary Hospital, Principal Investigator, Clinical Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L20-209
Record Dates: First submitted 2022-08-03; First posted 2022-08-09 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: MDR-TB; Immunotherapy
Keywords: MDR-TB；Immunotherapy；
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Drug Combinations; Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vγ2Vδ2 T lymphocyte-based immunotherapy +Treatment regimens for MDR-TB (Experimental): Treatment was based on the principles of the WHO guidelines for the treatment of drug-resistant tuberculosis, with the addition of immunotherapy：zoledronic acid and recombinant human interleukin 2
  Interventions: Drug: Vγ2Vδ2 T lymphocyte-based immunotherapy; Drug: Treatment regimens for MDR-TB
- Treatment regimens for MDR-TB (Active Comparator): Treatment regimens was based on the principles of the WHO guidelines for the treatment of drug-resistant tuberculosis.
  Interventions: Drug: Treatment regimens for MDR-TB

INTERVENTIONS:
Drug: Vγ2Vδ2 T lymphocyte-based immunotherapy — Intravenous injection of zoledronic acid, followed by a subcutaneous injection recombinant human interleukin. Zoledronic acid was administered 3 times and recombinant human interleukin was administered 10 times for a total of 6 months.
  Other Names: Drug combination (zoledronic acid/interleukin 2)
  Arms: Vγ2Vδ2 T lymphocyte-based immunotherapy +Treatment regimens for MDR-TB
Drug: Treatment regimens for MDR-TB — Treatment regimens was based on the principles of the WHO guidelines for the treatment of drug-resistant tuberculosis.
  Other Names: Treatment regimen for MDR-TB using WHO guidelines

SUMMARY:
A Exploratory Study of drug combination (zoledronic acid/interleukin 2) that specifically amplifies Vγ2Vδ2 T cells in combination with anti-tuberculosis chemotherapy for the treatment of MDR-TB.

DETAILED DESCRIPTION:
The emergence and prevalence of drug-resistant TB in recent years has made TB control more challenging, and MDR-TB is more serious type of drug-resistance TB with a cure rate of just over half, even with the latest treatment regimens. Treatment modalities other than drugs should be considered for patients with drug-resistant TB who have poor treatment efficacy, for patients with drug-resistant TB who are unresponsive to treatment, and for other patients for whom an effective treatment regimen cannot be composed.

The human immune system plays an important role in the infection, development, treatment and regression of tuberculosis.Mtb is an intracellularly parasitic bacterium that evades host immune clearance.Immunotherapy for TB can kill intracellularly parasitic Mycobacterium tuberculosis, including drug-resistant Mycobacterium tuberculosis, by inducing a host-specific immune response.The combination of antituberculosis chemotherapy and immunotherapy has the potential to open up new avenues for the treatment of multidrug-resistant TB.

In recent years, several studies by our team and others addressing host immune mechanisms have shown that γδ T cells play an important role in the fight against TB infection.Vγ2Vδ2 T cells (also known as Vγ9Vδ2 T cells) are a specific subset of γδ T cells, the only γδ T cells capable of recognizing TB phosphoantigens, and are found only in human and non-human primates.

Our previous study demonstrated that zoledronic acid, an anti-osteoporotic and osteoprotective drug, induced the production of endogenous ligands for Vγ2Vδ2T cells and activated Vγ2Vδ2T cells. Zoledronic acid in combination with interleukin 2 can significantly expand Vγ2Vδ2T cells, and the expanded Vγ2Vδ2T cells can effectively kill intracellular parasitic Mycobacterium tuberculosis, it can also promote the production of more anti-tuberculosis effectors by Vγ2Vδ2T cells and widely stimulate the production of functional cytokines by CD4 and CD8 T cells.

The primate experiments conducted by our team in the ABSL-III laboratory of Wuhan University demonstrated that phosphoantigen/interleukin 2 in a macaque model of tuberculosis infection induced lung phosphoantigen-specific Vγ2Vδ2 T cell expansion and migration, reduced Mycobacterium tuberculosis load in vivo, and effectively improved immune resistance to tuberculosis lung necrosis, demonstrating that targeted Vγ2Vδ2 T cell Immunotherapy of Vγ2Vδ2 T cells has a significant therapeutic effect on TB infection in monkeys , and is also safe for use in macaques. Accordingly, the investigators propose a drug combination (zoledronic acid/interleukin 2) that specifically amplifies Vγ2Vδ2 T cells in combination with anti-tuberculosis chemotherapy for the treatment of multidrug-resistant tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* RR-TB/MDR-TB (resistant to at least isoniazid and rifampicin).
* Poor efficacy of the original treatment regimen or no response to treatment or less than 4 effective drugs.

Exclusion Criteria:

* Immunosuppression due to co-morbidities, such as immune system disorders, tumors, etc.
* Test confirms poor response to ZOL and IL-2 stimulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2027-08-03 (Estimated)

PRIMARY OUTCOMES:
Sputum smear and culture negative conversion | Through study completion, an average of 24 months.
  Sputum smear microscopy, bacterial culture. Bacterial culture was performed via a mycobacterial growth indicator tube (MGIT) using the BACTEC MGIT 960 system.

SECONDARY OUTCOMES:
Radiographic changes | Through study completion, an average of 24 months.
  Radiographic changes after treatment compared to baseline.Outcomes were defined as unchanged or deteriorated; ecovered; improved based on radiological findings compared to baseline.

OTHER OUTCOMES:
Treatment outcome | Through study completion, an average of 24 months.
  Treatment outcome assessed at the end of the treatment course according to the new definitions released by the WHO.Classified as Treatment success (cure, treatment completion); Treatment failure, Death, Loss, Inconclusive.
Adverse reactions | Through study completion, an average of 24 months.
  Adverse reactions to drugs: Number of patients with Grade 3 or 4 Adverse Events，using a Modified Division of Acquired Immunodeficiency Syndrome National Institute of Allergy and Infectious Diseases [DAIDS] Scale of Adverse Event Reporting
Immunological indicators | Through study completion, an average of 24 months.
  The ability of Vγ2Vδ2 T cells to produce functional cytokines was analyzed. The results were enhanced/reduced cytokine production.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Pulmonary Hospital, Shanghai, China, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No